CLINICAL TRIAL: NCT04191746
Title: BEST Critical Limb Ischemia (vCLI) Registry
Brief Title: BEST vCLI Registry
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00102178; 1R01HL141213-01 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-12-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with critical limb disease: This registry will collect data from participants with critical limb disease from Duke University and approximately 40 sites in North America.

SUMMARY:
For subjects with critical limb ischemia, identify patient, physician/hospital, and geographic factors associated with variations in treatment strategies; compare treatments and outcomes, including quality of life, cost and cost effectiveness, at 6, 12 months.

DETAILED DESCRIPTION:
The study will be a prospective multicenter registry evaluating the real world therapeutic strategies, clinical outcomes, and costs associated with patients presenting with critical limb ischemia.

Population: Patients over age 18 presenting with critical limb ischemia After initial enrollment at 40 study sites throughout the US. participants will complete follow-up 6 months and 12 months via call center telephone calls.

The study plan calls for enrollment of approximately 1,200 participants throughout the US that will then have 12 month followup that includes collection of medications, hospitalizations for collection of events.Additionally, the BEST-CLI trial will be gathering quality of life data and cost data using similar instruments, thus providing an opportunity for comparison between cost and quality of life analyses in a clinical trial versus in a real-world registry and collection of Quality of Life using validated instruments: EQ-5D, VASQOL, SF-12.and bill review to determine economic impact of disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* age 18 years or older
* Infrainguinal peripheral artery disease (occlusive disease of the arteries below the inguinal ligament)
* Critical limb ischemia, defined as arterial insufficiency with gangrene, non-healing ischemic ulcer, or rest pain consistent with Rutherford categories 4-6
* Documented consideration for enrollment in the BEST-CLI Trial with documented failure to meet inclusion / exclusion criteria. Phase ll After BEST CLI official enrollment ends, this inclusion criteria will be removed.
* Willingness to comply with vCLI protocol, attend follow-up appointments, complete all study assessments, and provide written informed consent.

Exclusion Criteria:

* Presence of a popliteal aneurysm (> 2 cm) in the index limb
* Life expectancy of less than 2 years due to reasons other than peripheral artery disease
* Active vasculitis, Buerger's disease, or acute limb-threatening ischemia
* Current chemotherapy or radiation therapy
* Pregnancy or lactation
* Administration of an investigational drug for peripheral artery disease within 30 days of randomization
* Participation in a clinical trial (except observational studies) within the previous 30 days
* Prior enrollment or randomization into the BEST-CLI trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with critical limb ischemia Phase I: While the BEST-CLI Trial is actively enrolling, the BEST-Registry will only enroll patients who first screen fail from BEST-CLI.
  Phase II: After BEST-CLI officially finishes enrollment, screen failure for BEST-CLI will no longer be required for enrollment into the BEST-Registry
  1200 patients, across approximately 40 sites participating in BEST-CLI clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with major adverse limb events (MALE) as measured by patient reports (verified by medical records) | 6 months
  Number of participants in the registry with major limb events as reported by participants and confirmed by medical records
Percentage of participants with major adverse limb events (MALE) as measured by patient reports (verified by medical records) | 12 months
  Number of participants in the registry with major limb events as reported by participants and confirmed by medical records

SECONDARY OUTCOMES:
Number of participants that died within 30 days of index procedure | 30 days
  Collect composite of MALE or perioperative death within 30 days of index procedure using patient/proxy information qualified by medical records.
Number of participants with amputation free survival as measured by patient report/verified by medical record review | 6 months
  Interviews completed at 6 months with participants that note no hospitalization for amputation and verified by medical records
Number of participants with amputation free survival as measured by patient report/verified by medical record review | 12 months
  Interviews completed at 12 months with participants that note no hospitalization for amputation and verified by medical records
Number of participants that did not have secondary interventions in index leg as measured by patient report/verified by medical record review | 6 months
  At 6 month visit, the number of participants that did not report additional procedures such as surgery or angiography.in the affected leg
Number of participants that did not have secondary interventions in index leg as measured by patient report/verified by medical record review | 12 months
  At 12 month visit, the number of participants that did not report additional procedures such as surgery or angiography.in the affected leg
Number of interventions per limb as measured by patient report/verified by medical record review | 6 months
  Interventions consist of need to be hospitalized for a form of revascularization
Number of interventions per limb as measured by patient report/verified by medical record review | 12 months
  Interventions consist of need to be hospitalized for a form of revascularization
Number of participants that did not have limb revascularization failure as measured by patient report/verified by medical record review | 6 months
  Limb revascularization failure is loss of circulation to the limb that has procedural revascularization previously performed that is non functioning
Number of participants that did not have limb revascularization failure as measured by patient report/verified by medical record review | 12 months
  Limb revascularization failure is loss of circulation to the limb that has procedural revascularization previously performed that is non functioning
Number of participants who did not have a myocardial infarction as measured by patient report/verified by medical record review | 6 months
  Number of participants that answered no to the question "Was your hospitalization for a Heart Attack(MI) at 6 months verified by medical record.
Number of participants who did not have a myocardial infarction as measured by patient report/verified by medical record review | 12 months
  Number of participants that answered no to the question "Was your hospitalization for a Heart Attack(MI) at 12 months verified by medical record.
Number of participants who did not have a stroke while in the registry as measured by patient report/verified by medical record review | 6 months
  Stroke is inclusive of a cerebral vascular including a ischemic, hemorrhagic or a TIA event.
Number of participants who did not have a stroke while in the registry as measured by patient report/verified by medical record review | 12 months
  Stroke is inclusive of a cerebral vascular including a ischemic, hemorhagic or a TIA event.
Number of participants that did not have a periprocedural (30 day) major adverse cardiac events as measured by patient report/verified by medical record review | 6 months
  Events that occur during a revascularization procedure including cardiovascular events such as Myocardial Infarction and stoke.
Quality of life as measure by the validated QOL tool called the EuroQol that will be administered throughout the study | Baseline
  The EuroQol is a 6 question validated instrument that asks questions regarding mobility, self care, usual activities, pain/discomfort and anxiety and depression. I also includes a 0-100 scale regarding participants assessment of health.
Quality of life as measure by the validated QOL tool called the EuroQol that will be administered throughout the study | 6 month
  The EuroQol is a 6 question validated instrument that asks questions regarding mobility, self care, usual activities, pain/discomfort and anxiety and depression. I also includes a 0-100 scale regarding participants assessment of health.
Quality of life as measure by the validated QOL tool (EuroQol) that will be administered throughout the study | 12 month
  The EuroQol is a 6 question validated instrument that asks questions regarding mobility, self care, usual activities, pain/discomfort and anxiety and depression with a range of 5 answers. I also includes a 0-100 scale regarding participants assessment of health.
Quality of life as measured by the the SF-12 instrument that will be administered throughout the study | Baseline
  The SF-12 Health Survey is a shorter version of the SF-36 Health Survey that uses 12 questions to measure functional health and well-being from the patient's point of view
Quality of life as measured by the the SF-12 instrument that will be administered throughout the study | 6 months
  The SF-12 Health Survey is a shorter version of the SF-36 Health Survey that uses 12 questions to measure functional health and well-being from the patient's point of view
Quality of life as measured by the the SF-12 instrument that will be administered throughout the study | 12 months
  The SF-12 Health Survey is a shorter version of the SF-36 Health Survey that uses 12 questions to measure functional health and well-being from the patient's point of view

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Patel, MD, Principal Investigator — Duke University; Sreekanth Vemulapalli, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No